CLINICAL TRIAL: NCT02761005
Title: Eradication of H. Pylori With the Regimen Individualized Susceptibility of H. Pylori to Clarithromycin Determined by the Mutation of 23S rRNA of H. Pylori
Brief Title: Eradication of H. Pylori Therapy Individualized by the Mutation of 23S rRNA of H. Pylori
Acronym: EHR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Takahisa Furuta, Professor, Hamamatsu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hp23SrRNA
Record Dates: First submitted 2016-04-25; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: H. Pylori Infection
Keywords: Eradication therapy; Mutation of 23S rRNA of H. pylori; Personalized therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 23S rRNA wt (Experimental): As the 23S rRNA mutation guided selection of antimicrobial agent, patients infected with strains without mutation of 23S rRNA are assigned to this arm. In this arm, they are treated with vonoprazan 20 mg bid, amoxicillin 750 mg bid and clarithromycin 200 mg bid for 1 week for the eradication of H. pylori.
  Interventions: Drug: Eradication of H. pylori
- 23S rRNA mutation (Experimental): As the 23S rRNA mutation guided selection of antimicrobial agent, patients infected with strains with mutation of 23S rRNA are assigned to this arm. In this arm, they are treated with vonoprazan 20 mg bid, amoxicillin 750 mg bid and metronidazole 250 mg bid for 1 week for the eradication of H. pylori,
  Interventions: Drug: Eradication of H. pylori

INTERVENTIONS:
Drug: Eradication of H. pylori — For the eradication of H. pylori, patients diagnosed to be infected with strain with mutation of 23S rRNA, their H. pylori strains are considered to be resistant to clarithromycin. Then, they are treated with vonoprazan 40 mg, metronidazole 500 mg and amoxicillin 1500 mg for 1 week. Patients diagnosed to be infected with strain without mutation of 23S rRNA, their H. pylori strains are considered to be resistant to clarithromycin. Then, they are treated with vonoprazan 40 mg, clarithromycin 400 mg and amoxicillin 1500 mg for 1 week.
  Other Names: Eradication regimen for H. pylori based on SNPs of 23S RNA; Tailored eradication based on genetics

SUMMARY:
Patients infected with H. pylori are treated with the individualized regimen which is based on the mutation of 23S rRNA of H. pylori.

DETAILED DESCRIPTION:
Patients infected with H. pylori undergo the gastroscopy. During the gastroscopy, gastric mucus samples are collected, from which DNA is extracted. The DNA samples are subjected the full-auto SNP analyzer and the from A to G mutation of 23s rRNA of H. pylori at the positions of 2142 and 2143 is measured. When the mutation is detected, patients are diagnosed to be infected with clarithromycin-resistant strains of H. pylori and therefore, treated with the triple therapy with vonoprazan 20 mg bid + amoxicillin 750 mg bid + metronidazole 250 mg bid for 1 week. When the mutation is not detected, patients are considered to be infected with clarithromycin-sensitive strains of H. pylori and therefore, treated with the triple therapy with vonoprazan 20 mg bid + amoxicillin 750 mg bid + clarithromycin 200 mg bid for 1 week. The success or failure of eradication was determined based on the 13C-urea breath test performed 1 month after the therapy. The total eradication rates with this strategy was compared with that by the standard regimen in Japan performed in the same period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with H. pylori are invited to the study.
* Patients not allergic to the any of the drugs used for eradication of H. pylori.
* Patients who has agreed to participate to the study.

Exclusion Criteria:

* Patients allergic to the any of the drugs used for eradication of H. pylori.
* Patients who do not agree to the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Eradication rates | Eradication of H. pylori is measured 1 month after the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Takahisa Furuta, MD, PhD, Principal Investigator — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan

IPD SHARING:
Plan to Share IPD: No
The data obtained with this study are restricted in our hospital.